CLINICAL TRIAL: NCT00917384
Title: A Phase 3, Randomized, Double-Blinded Study of IMC-1121B and Best Supportive Care (BSC) Versus Placebo and BSC in the Treatment of Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma Following Disease Progression on First-Line Platinum- or Fluoropyrimidine-Containing Combination Therapy
Brief Title: Study of IMC-1121B (Ramucirumab) With Best Supportive Care in Participants With Gastric Cancer and Adenocarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13893; 2008-005964-15 (Registry Identifier: MHRA); CP12-0715 (Other: ImClone Systems); I4T-IE-JVBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer; Adenocarcinoma
Keywords: IMC-1121B; Monoclonal antibody (MAb); Vascular endothelial growth factor (VEGF); Human vascular endothelial growth factor receptor-2 (VEGFR-2); Platinum resistant; platinum refractory; Gastric; Gastroesophageal Junction Adenocarcinoma; metastatic; Angiogenesis
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — Ramucirumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ramucirumab (Experimental): Participants receive ramucirumab, administered via intravenous infusion every 2 weeks at a dose of 8 milligrams/kilogram (mg/kg), and best supportive care (BSC) as determined appropriate by the investigator(s). Treatment will continue until there is evidence of progressive disease (PD), the development of unacceptable toxicity, protocol noncompliance, or withdrawal of consent.
  Interventions: Biological: ramucirumab; Other: Best Supportive Care (BSC)
- Placebo (Placebo Comparator): Participants receive injection for intravenous infusion every 2 weeks plus BSC as determined appropriate by the investigator(s). Because investigators and ancillary medical personnel will be blinded as to assignment to active therapy versus placebo, the volume of placebo to be administered will be calculated as if it were active product with a dose of 8 mg/kg. Treatment will continue until there is evidence of PD, the development of unacceptable toxicity, protocol noncompliance, or withdrawal of consent.
  Interventions: Drug: Placebo; Other: Best Supportive Care (BSC)

INTERVENTIONS:
Biological: ramucirumab — Administered via intravenous infusion every 2 weeks at a dose of 8 mg/kg
  Other Names: IMC-1121B; LY3009806
  Arms: ramucirumab
Drug: Placebo — Placebo comparator for ramucirumab 8 mg/kg as intravenous infusion every 2 weeks
  Arms: Placebo
Other: Best Supportive Care (BSC) — BSC as determined appropriate by the investigator(s). BSC may include but are not limited to antiemetic agents, opiate and nonopiate analgesic agents, appetite stimulants, and granulocyte and erythroid growth factors.

SUMMARY:
The purpose of this study is to gather information about the use of an investigational drug called Ramucirumab in adenocarcinomas of the stomach or gastroesophageal junction.

DETAILED DESCRIPTION:
Placebo-controlled, multicenter Phase 3 study of participants with metastatic gastric cancer [including adenocarcinomas of the gastroesophageal junction (GEJ)] and disease progression on standard first-line chemotherapeutic regimens. Participants will be randomized on a 2:1 basis to receive best supportive care plus ramucirumab administered every 2 weeks or best supportive care plus placebo administered every 2 weeks, respectively. Participants will undergo radiographic assessment of disease status every 6 weeks. Participant will be treated until there is evidence of progressive disease, toxicity requiring cessation, withdrawal of consent, or until other withdrawal criteria are met.

Approximately 348 participants, with histologically- or cytologically-confirmed, metastatic gastric or GEJ adenocarcinoma, and radiographically measurable disease as defined by the Response Evaluation Criteria in Solid Tumors or evaluable, nonmeasurable disease, will be randomized. Participants will be enrolled from approximately 250 study centers in North America, South America, Central America, Asia, Australia, New Zealand, and Europe.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed gastric carcinoma, including gastric adenocarcinoma or GEJ adenocarcinoma
* Metastatic disease or locally recurrent, unresectable disease with measurable lymph node metastases
* Measurable disease and/or evaluable disease. Measurable disease is defined as at least one unidimensionally-measurable target lesion [≥ 2 centimeter (cm) with conventional techniques or ≥ 1 cm by spiral computed tomography (CT)], as defined by Response using Response Evaluation Criteria in Solid Tumors (RECIST).

Examples of evaluable, nonmeasurable disease include gastric, peritoneal, or mesenteric thickening in areas of known disease, or peritoneal nodules that are too small to be considered measurable by RECIST

* Experienced disease progression during or within 4 months after the last dose of first-line therapy for metastatic disease, or during or within 6 months after the last dose of adjuvant therapy
* Disease is not amenable to potentially curative resection
* Participant is ≥ 18 years of age
* Participant has a life expectancy of ≥ 12 weeks
* Participant resolution to Grade ≤ 1 (or to Grade ≤ 2 in the case of neuropathy) by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3.0, of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy (with the exception of alopecia)
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0-1
* The participant has adequate hepatic function as defined by a total bilirubin ≤ 1.5 milligrams/deciliter (mg/dL) [25.65 micromole/liter (µmol/L)], and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x the upper limit of normal (ULN) [or 5.0 x the ULN in the setting of liver metastases]
* The participant has adequate renal function as defined by a serum creatinine ≤ 1.5 x the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥ 40 milliliters/minute (mL/min) (that is, if serum creatinine is > 1.5 x the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed)
* The participant's urinary protein is ≤ 1+ on dipstick or routine urinalysis ([UA]; if urine dipstick or routine analysis is ≥ 2+, a 24-hour urine collection for protein must demonstrate < 1000 milligrams (mg) of protein in 24 hours to allow participation in the study)
* The participant has adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥ 1000 microliters (µL), hemoglobin ≥ 9 grams/deciliter (g/dL) [5.58 millimoles/liter (mmol/L)], and platelets ≥ 100,000/µL
* The participant must have adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5 and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Participant on anticoagulation therapy with unresected primary tumors or local tumor recurrence following resection are not eligible
* If the participant has received prior anthracycline therapy as part of his or her first-line regimen, the participant is able to engage in ordinary physical activity without significant fatigue or dyspnea
* Because the teratogenicity of IMC-1121B is not known, the participant, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods)
* Female participant of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization
* Able to provide informed written consent and is amenable to compliance with protocol schedules and testing

Exclusion Criteria:

* Documented and/or symptomatic brain or leptomeningeal metastases
* Experienced any Grade 3-4 gastrointestinal bleeding within 3 months prior to randomization
* Experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to randomization
* Ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the investigator
* Ongoing or active psychiatric illness or social situation that would limit compliance with study requirements
* Uncontrolled or poorly-controlled hypertension despite standard medical management
* Participant has a serious or nonhealing wound, ulcer, or bone fracture
* Received chemotherapy, radiotherapy, immunotherapy, or targeted therapy for gastric cancer within 2 weeks prior to randomization
* Received any investigational therapy within 30 days prior to randomization
* Undergone major surgery within 28 days prior to randomization, or subcutaneous venous access device placement within 7 days prior to randomization
* Received prior therapy with an agent that directly inhibits vascular endothelial growth factor (VEGF) or VEGF receptor 2 (R-2) activity (including bevacizumab), or any antiangiogenic agent
* Receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use [maximum dose 325 milligram/day (mg/day)] is permitted
* Participant has elective or planned major surgery to be performed during the course of the clinical trial
* Participant has a known allergy to any of the treatment components
* Pregnant or lactating
* Known to be positive for infection with the human immunodeficiency virus
* Known alcohol or drug dependency
* Participant has a concurrent active malignancy other than adequately-treated nonmelanomatous skin cancer, other noninvasive carcinoma, or in situ neoplasm. A participant with previous history of malignancy is eligible, provided that he/she has been free of disease for > 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (135):
- United States (14):
  - ImClone Investigational Site, Bakersfield, California
  - ImClone Investigational Site, La Jolla, California
  - ImClone Investigational Site, Redlands, California
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, New Orleans, Louisiana
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, Omaha, Nebraska
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, West Reading, Pennsylvania
  - ImClone Investigational Site, Providence, Rhode Island
  - ImClone Investigational Site, Charleston, South Carolina
  - ImClone Investigational Site, Knoxville, Tennessee
  - ImClone Investigational Site, Memphis, Tennessee
  - ImClone Investigational Site, Houston, Texas
- Argentina (5):
  - ImClone Investigational Site, Buenos Aires
  - ImClone Investigational Site, Capital Federal
  - ImClone Investigational Site, Ciudada Autonoma
  - ImClone Investigational Site, Córdoba
  - ImClone Investigational Site, Rosario
- Australia (7):
  - ImClone Investigational Site, Wodonga, New South Wales
  - ImClone Investigational Site, Hobart, Tasmania
  - ImClone Investigational Site, East Melbourne, Victoria
  - ImClone Investigational Site, Perth, Western Australia
  - ImClone Investigational Site, Bedford Park
  - ImClone Investigational Site, St Leonards
  - ImClone Investigational Site, Woodville
- ImClone Investigational Site, Sarajevo, Bosnia and Herzegovina
- Brazil (11):
  - ImClone Investigational Site, Barretos
  - ImClone Investigational Site, Belo Horizonte
  - ImClone Investigational Site, Brasília
  - ImClone Investigational Site, Curitiba
  - ImClone Investigational Site, Florianópolis
  - ImClone Investigational Site, Ijuí
  - ImClone Investigational Site, Lajeados
  - ImClone Investigational Site, Londrina
  - ImClone Investigational Site, Passo Fundo
  - ImClone Investigational Site, Porto Alegre
  - ImClone Investigational Site, São Paulo
- Canada (3):
  - ImClone Investigational Site, Edmonton, Alberta
  - ImClone Investigational Site, Montreal, Quebec
  - ImClone Investigational Site, Sherbrooke, Quebec
- Chile (3):
  - ImClone Investigational Site, Concepción
  - ImClone Investigational Site, La Serena
  - ImClone Investigational Site, Santiago
- ImClone Investigational Site, Montería, Colombia
- Croatia (4):
  - ImClone Investigational Site, Osijek
  - ImClone Investigational Site, Pula
  - ImClone Investigational Site, Slavonski Brod
  - ImClone Investigational Site, Zagreb
- Czechia (8):
  - ImClone Investigational Site, Brno
  - ImClone Investigational Site, Hradec Králové
  - ImClone Investigational Site, Liberec
  - ImClone Investigational Site, Nová Ves pod Pleší
  - ImClone Investigational Site, Olomouc
  - ImClone Investigational Site, Pardubice
  - ImClone Investigational Site, Prague
  - ImClone Investigational Site, Příbram
- Egypt (2):
  - ImClone Investigational Site, Alexandria
  - ImClone Investigational Site, Cairo
- ImClone Investigational Site, Guatemala City, Guatemala
- India (21):
  - ImClone Investigational Site, Hyderabad, ANDH PRAD
  - ImClone Investigational Site, Bangalore, Karna
  - ImClone Investigational Site, Kochi, Kerala
  - ImClone Investigational Site, Thiruvananthapuram, Kerala
  - ImClone Investigational Site, Trivandrum, Kerala
  - ImClone Investigational Site, Chennai, Kilpauk
  - ImClone Investigational Site, Bhopal, MADH PRAD
  - ImClone Investigational Site, Indore, MADH PRAD
  - ImClone Investigational Site, Mumbai, Mahara
  - ImClone Investigational Site, Nashik, Mahara
  - ImClone Investigational Site, Pune, Mahara
  - ImClone Investigational Site, New Delhi, National Capital Territory of Delhi
  - ImClone Investigational Site, Chennai, Tamil Nadu
  - ImClone Investigational Site, Kolkata, West Bengal
  - ImClone Investigational Site, Bangalore
  - ImClone Investigational Site, Chennai
  - ImClone Investigational Site, Hyderabad
  - ImClone Investigational Site, Kolkata
  - ImClone Investigational Site, Mumbai
  - ImClone Investigational Site, Pune
  - ImClone Investigational Site, West Bengal
- Indonesia (3):
  - ImClone Investigational Site, Jakarta
  - ImClone Investigational Site, Sumatera Utara
  - ImClone Investigational Site, West Java
- Italy (12):
  - ImClone Investigational Site, Aviano
  - ImClone Investigational Site, Bologna
  - ImClone Investigational Site, Brescia
  - ImClone Investigational Site, Cremona
  - ImClone Investigational Site, Lido di Camaiore
  - ImClone Investigational Site, Lucca
  - ImClone Investigational Site, Meldola
  - ImClone Investigational Site, Mirano
  - ImClone Investigational Site, Noale
  - ImClone Investigational Site, Potenza
  - ImClone Investigational Site, Rimini
  - ImClone Investigational Site, Udine
- ImClone Investigational Site, Beirut, Lebanon
- ImClone Investigational Site, Floriana, Malta
- ImClone Investigational Site, Aguascelientes, Mexico
- ImClone Investigational Site, Christchurch, New Zealand
- Philippines (2):
  - ImClone Investigational Site, Cebu City
  - ImClone Investigational Site, Pasig
- Poland (3):
  - ImClone Investigational Site, Gdansk
  - ImClone Investigational Site, Krakow
  - ImClone Investigational Site, Olsztyn
- Romania (3):
  - ImClone Investigational Site, Baia Mare
  - ImClone Investigational Site, Cluj-Napoca
  - ImClone Investigational Site, Suceava
- Russia (5):
  - ImClone Investigational Site, Chelyabinsk
  - ImClone Investigational Site, Kursk
  - ImClone Investigational Site, Moscow
  - ImClone Investigational Site, Pyatigorsk
  - ImClone Investigational Site, Saint Petersburg
- ImClone Investigational Site, Cape Town, South Africa
- ImClone Investigational Site, Seoul, South Korea
- Spain (6):
  - ImClone Investigational Site, Alcorcón
  - ImClone Investigational Site, Barcelona
  - ImClone Investigational Site, Elche
  - ImClone Investigational Site, Madrid
  - ImClone Investigational Site, Santander
  - ImClone Investigational Site, Seville
- Taiwan (3):
  - ImClone Investigational Site, Kaohsiung City
  - ImClone Investigational Site, Taichung County
  - ImClone Investigational Site, Taipei
- Thailand (3):
  - ImClone Investigational Site, Bangkok
  - ImClone Investigational Site, Chiang Mai
  - ImClone Investigational Site, Rajathevee District
- Turkey (Türkiye) (4):
  - ImClone Investigational Site, Adana
  - ImClone Investigational Site, Gaziantep
  - ImClone Investigational Site, Istanbul
  - ImClone Investigational Site, Izmir
- United Kingdom (4):
  - ImClone Investigational Site, Bebington, Wirral
  - ImClone Investigational Site, London
  - ImClone Investigational Site, Sutton
  - ImClone Investigational Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Chau I, Fuchs CS, Ohtsu A, Barzi A, Liepa AM, Cui ZL, Hsu Y, Al-Batran SE. Association of quality of life with disease characteristics and treatment outcomes in patients with advanced gastric cancer: Exploratory analysis of RAINBOW and REGARD phase III trials. Eur J Cancer. 2019 Jan;107:115-123. doi: 10.1016/j.ejca.2018.11.013. Epub 2018 Dec 14. PMID 30557792
- [Derived] Tabernero J, Ohtsu A, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Ajani JA, Tomasek J, Safran H, Chandrawansa K, Hsu Y, Heathman M, Khan A, Ni L, Melemed AS, Gao L, Ferry D, Fuchs CS. Exposure-Response Analyses of Ramucirumab from Two Randomized, Phase III Trials of Second-line Treatment for Advanced Gastric or Gastroesophageal Junction Cancer. Mol Cancer Ther. 2017 Oct;16(10):2215-2222. doi: 10.1158/1535-7163.MCT-16-0895. Epub 2017 Jul 17. PMID 28716815
- [Derived] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Participant Flow participants who completed were those who died due to any cause or were alive and on study at conclusion but off treatment.
Groups:
- IMC-1121B (Ramucirumab ): Participants received IMC-1121B (ramucirumab), administered via intravenous infusion every 2 weeks at a dose of 8 milligrams/kilogram (mg/kg), plus best supportive care (BSC) as determined appropriate by the investigator(s). Treatment continued until there was evidence of progressive disease (PD), the development of unacceptable toxicity, protocol noncompliance, or withdrawal of consent.
- Placebo: Participants received placebo by intravenous infusion every 2 weeks plus BSC as determined appropriate by the investigator(s). Because investigators and ancillary medical personnel were blinded as to assignment to active therapy versus placebo, the volume of placebo administered was calculated as if it were active product with a dose of 8 mg/kg. Treatment continued until there was evidence of PD, the development of unacceptable toxicity, protocol noncompliance, or withdrawal of consent.
Period: Overall Study
Arm/Group | IMC-1121B (Ramucirumab ) | Placebo
Started | 238 | 117
Received at Least 1 Dose of Study Drug | 236 | 115
Completed | 224 | 113
Not Completed | 14 | 4
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 10 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- IMC-1121B (Ramucirumab): Participants received IMC-1121B (ramucirumab), administered via intravenous infusion every 2 weeks at a dose of 8 milligrams/kilogram (mg/kg), plus best supportive care (BSC) as determined by the investigator(s). Treatment continued until there was evidence of progressive disease (PD), the development of unacceptable toxicity, protocol noncompliance, or withdrawal of consent.
- Placebo: Participants received placebo by intravenous infusion every 2 weeks plus best supportive care as determined appropriate by the investigator(s). Because investigators and ancillary medical personnel were blinded as to assignment to active therapy versus placebo, the volume of placebo administered was calculated as if it were active product with a dose of 8 mg/kg. Treatment continued until there was evidence of PD, the development of unacceptable toxicity, protocol noncompliance, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | IMC-1121B (Ramucirumab) | Placebo | Total
Number analyzed (Participants) | 238 | 117 | 355
Age, Continuous [Median (Full Range); unit: years] | 60.0 [30 to 86] | 60.0 [24 to 87] | 60.0 [24 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 38 | 107
  Male | 169 | 79 | 248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 19 | 60
  Not Hispanic or Latino | 197 | 98 | 295
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 4 | 2 | 6
  Australia | 8 | 4 | 12
  Bosnia and Herzegovina | 1 | 3 | 4
  Brazil | 24 | 14 | 38
  Canada | 8 | 2 | 10
  Chile | 1 | 1 | 2
  Colombia | 2 | 1 | 3
  Czech Republic | 24 | 13 | 37
  Egypt | 1 | 0 | 1
  Spain | 12 | 4 | 16
  United Kingdom | 13 | 4 | 17
  Guatemala | 6 | 2 | 8
  Croatia | 7 | 0 | 7
  Indonesia | 2 | 1 | 3
  India | 16 | 8 | 24
  Italy | 23 | 11 | 34
  Korea, Republic of | 11 | 6 | 17
  Lebanon | 1 | 0 | 1
  Malta | 2 | 3 | 5
  New Zealand | 1 | 1 | 2
  Philippines | 1 | 1 | 2
  Poland | 9 | 4 | 13
  Romania | 13 | 4 | 17
  Russian Federation | 14 | 8 | 22
  Thailand | 1 | 0 | 1
  Turkey | 5 | 1 | 6
  Taiwan | 3 | 0 | 3
  United States | 25 | 18 | 43
  South Africa | 0 | 1 | 1
Race [Number; unit: participants]
  White | 181 | 91 | 272
  Asian | 39 | 17 | 56
  Black | 4 | 2 | 6
  Other | 14 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death from any cause. Participants who were alive at the date of data cut-off or who were lost to follow-up were censored on the last date the participant was known to be alive
Time Frame: Randomization up to 28 months post-randomization
Population: Intent-to-treat population: all randomized participants. Censored participants: ramucirumab=59, placebo=18.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Number analyzed (Participants) | 238 | 117
months | 5.2 [4.4 to 5.7] | 3.8 [2.8 to 4.7]
Statistical Analysis 1: Comparison: IMC-1121B (Ramucirumab) vs Placebo; Test type: Superiority or Other; p = 0.0473, Stratified Log-Rank Test; Stratified Log-Rank Test and HR stratified by randomization strata (weight loss over the prior 3 months, primary tumor site and geographical region); Hazard Ratio (HR) = 0.776, 95% CI [0.603 to 0.998]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from date of randomization until date of objectively determined progressive disease (PD) or death due to any cause, whichever is first. Participants alive and without PD were censored at the time of last adequate objective tumor assessment (that is, response other than unevaluable).
Time Frame: Randomization up to 17 months
Population: Intent-to-treat population: all randomized participants. Censored participants: ramucirumab=39, placebo=9.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Number analyzed (Participants) | 238 | 117
months | 2.1 [1.5 to 2.7] | 1.3 [1.3 to 1.4]
Statistical Analysis 1: Comparison: IMC-1121B (Ramucirumab) vs Placebo; Test type: Superiority or Other; p < 0.0001, Stratified Log-Rank Test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.483, 95% CI 2-sided [0.376 to 0.620]

3. Secondary Outcome: Percentage of Participants Who Are Progression-Free at Week 12 (PFS Rate)
Description: The percentage of participants alive and progression-free 12 weeks after randomization. Progression-free survival (PFS) is defined as the time from the date of randomization until the date of objectively determined progressive disease (PD) or death due to any cause whichever comes first. Participants alive and without PD were censored at the time of the last adequate objective tumor assessment.
Time Frame: Week 12 post-randomization
Population: Intent-to-treat population: all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Number analyzed (Participants) | 238 | 117
percentage of participants | 40.1 [33.6 to 46.4] | 15.8 [9.7 to 23.3]
Statistical Analysis 1: Comparison: IMC-1121B (Ramucirumab) vs Placebo; Test type: Superiority or Other; p < 0.0001, Normal Approximation; Difference Between Arms = 24.2, 95% CI 2-sided [14.9 to 33.6]

4. Secondary Outcome: Percentage of Participants With Objective Response (Objective Response Rate [ORR])
Description: ORR is equal to the percentage of participants achieving a best overall response of complete response (CR) or partial response (PR). CR and PR were defined using the Response Evaluation Criteria in Solid Tumors (RECIST v1.0). CR is defined as the disappearance of all target and non-target lesions, no appearance of new lesions and confirmed at the consecutive tumor assessment. PR is defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, no appearance of new lesions and confirmed at a subsequent tumor assessment.
Time Frame: Randomization up to 17 months post-randomization
Population: Intent-to-treat population: all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Number analyzed (Participants) | 238 | 117
percentage of participants | 3.4 [1.5 to 6.5] | 2.6 [0.5 to 7.3]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is the interval from date of initial documented response (complete response [CR] or partial response [PR]) to first documented date of disease progression (PD) or death as a result of any cause. CR and PR were defined using the Response Evaluation Criteria in Solid Tumors (RECIST v1.0). CR is defined as the disappearance of all target and non-target lesions, no appearance of new lesions and confirmed at the consecutive tumor assessment. PR is defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, no appearance of new lesions and confirmed at a subsequent tumor assessment. Participants who did not relapse or die were censored at the time of the last adequate objective tumor assessment.
Time Frame: Randomization up to 17 months post-randomization
Population: Zero participants were analyzed. The number of all responders (participants with CR or PR) was too small for a meaningful analysis, as specified in the statistical analysis plan.
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Quality of Life (QoL) as Measured by the European Organisation for Research and Treatment of Cancer Questionnaire (EORTC-QLQ-C30)
Description: EORTC QLQ-C30 v3.0 is a self-administered questionnaire with multidimensional scales that measures 5 functional domains (physical, role, cognitive, emotional, and social), global health status, and symptom scales of fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation and diarrhea, and financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, higher scores represent a better level of functioning. For symptoms scales, higher scores represented a greater degree of symptoms. Best change from baseline results determined by Least Square (LS) mean estimated with randomization stratification factors and baseline value as continuous covariate.
Time Frame: Baseline up to Cycle 10 (18 weeks [1 cycle=2 weeks])
Population: All randomized participants with EORTC QLQ-C30 values at baseline and any point up to 18 weeks post-baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Number analyzed (Participants) | 114 | 26
units on a scale
  Global Health Status/QoL | 2.42 (2.99) | 0.80 (4.48)
  Physical Functioning | -6.26 (3.20) | -12.01 (4.82)
  Role Functioning | -4.32 (4.65) | -11.79 (6.99)
  Emotional Functioning | -1.61 (3.29) | -6.51 (4.92)
  Cognitive Functioning | -4.26 (2.63) | -10.94 (3.94)
  Social Functioning | -1.98 (3.90) | -1.37 (5.86)
  Fatigue | 3.16 (3.43) | 6.88 (5.16)
  Nausea and Vomiting | 1.77 (2.86) | 2.88 (4.32)
  Pain | 0.13 (3.61) | 3.85 (5.42)
  Dyspnea | -2.61 (3.35) | 3.51 (5.08)
  Insomnia | -7.47 (4.19) | -3.95 (6.28)
  Appetite Loss | -1.01 (4.60) | 7.16 (6.91)
  Constipation | 0.09 (3.79) | 7.94 (5.69)
  Diarrhea | -3.97 (1.64) | -5.49 (2.46)
  Financial Difficulties | -12.86 (3.78) | -2.39 (5.68)

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Clinically significant events were defined as serious adverse events (SAE) and other treatment-emergent non-serious adverse events (NSAE). A summary of SAEs and all other NSAEs is located in the Reported Adverse Event module.
Time Frame: Randomization up to 18 months
Population: Safety Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Number analyzed (Participants) | 236 | 115
participants
  Participants with SAE | 112 | 51
  Participants with ≥ 1 treatment emergent NSAE | 213 | 91

8. Secondary Outcome: Maximum Concentration (Cmax) of IMC-1121B
Description: Cmax was not analyzed as only pre-dose samples were collected.
Time Frame: 6 weeks post-randomization
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants Who Developed Antibodies Against IMC-1121B
Description: The number of participants who developed treatment emergent antibody responses to IMC-1121B after baseline.
Time Frame: Baseline, 12 Weeks
Population: Subset of the Safety Population: All randomized participants who received at least 1 dose of study drug and who had immunogenicity analysis performed.
Measure: Number; unit: participants
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Number analyzed (Participants) | 207 | 106
participants | 6 | 1

ADVERSE EVENTS:
Arm/Group | IMC-1121B (Ramucirumab) | Placebo
Serious Adverse Events (participants affected / at risk) | 112/236 | 51/115
Other Adverse Events (participants affected / at risk) | 213/236 | 91/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IMC-1121B (Ramucirumab) (N=236) | Placebo (N=115)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 2 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 6 (6) | 3 (4)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 3 (4)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (3)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 5 (5)
Asthenia (General disorders) | 0 (0) | 4 (4)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 5 (5) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 10 (10) | 8 (8)
Extravasation (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 4 (4) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 6 (6) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Drug dispensing error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 7 (8) | 1 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Underdose (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (7) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hyperammonaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal laceration (Reproductive system and breast disorders) | 1/67 (1) | 0/38 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Jejunostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Oesophageal stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-1121B (Ramucirumab) (N=236) | Placebo (N=115)
Anaemia (Blood and lymphatic system disorders) | 33 (41) | 16 (22)
Abdominal pain (Gastrointestinal disorders) | 40 (53) | 26 (36)
Abdominal pain upper (Gastrointestinal disorders) | 26 (35) | 5 (5)
Ascites (Gastrointestinal disorders) | 18 (23) | 8 (8)
Constipation (Gastrointestinal disorders) | 37 (53) | 24 (38)
Diarrhoea (Gastrointestinal disorders) | 35 (64) | 9 (12)
Dyspepsia (Gastrointestinal disorders) | 6 (8) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 23 (33) | 11 (22)
Nausea (Gastrointestinal disorders) | 45 (62) | 30 (44)
Vomiting (Gastrointestinal disorders) | 45 (70) | 26 (36)
Asthenia (General disorders) | 30 (60) | 16 (19)
Fatigue (General disorders) | 58 (90) | 28 (52)
Oedema peripheral (General disorders) | 21 (27) | 10 (11)
Weight decreased (Investigations) | 26 (34) | 11 (13)
Decreased appetite (Metabolism and nutrition disorders) | 55 (90) | 26 (39)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 (15) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (20) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (22) | 11 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (11) | 6 (11)
Dizziness (Nervous system disorders) | 4 (6) | 6 (7)
Dysgeusia (Nervous system disorders) | 7 (7) | 6 (9)
Headache (Nervous system disorders) | 21 (28) | 4 (4)
Insomnia (Psychiatric disorders) | 13 (14) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 15 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 1 (1)
Hypertension (Vascular disorders) | 35 (125) | 9 (31)
Hypotension (Vascular disorders) | 5 (6) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study completion or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.